CLINICAL TRIAL: NCT03633734
Title: Efficacy Evaluation of Sequential Treatment With Nab-paclitaxel Plus Gemcitabine and Modified Folfirinox in Metastatic Pancreatic Adenocarcinoma
Brief Title: Efficacy Evaluation of Sequential Treatment With AG and Modified Folfirinox in Metastatic Pancreatic Adenocarcinoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAHZJU-Y2018-058
Record Dates: First submitted 2018-08-14; First posted 2018-08-16 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Pancreatic Adenocarcinoma Metastatic; Chemotherapy Effect
Keywords: Pancreatic cancer; Pancreatic Adenocarcinoma; Gemcitabine; Nab-paclitaxel; Modified Folfirinox; Sequential treatment
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sequential treatment (Experimental): One cycle of sequential treatment lasts for 56 days.
  1. Stage 1(28 days): AG regimen. Nab-paclitaxel (Abraxane) 125mg/m^2 + gemcitabine 1000mg/m^2 (days 1, 8, 15, 28)
  2. Stage 2(28 days)：mFolfirinox regimen. Fluorouracil 2400 mg/m^2 continuous intravenous drip 46h + calcium folinate 400 mg/m^2 + irinotecan 135 mg/m^2 + oxaliplatin 68 mg/m^2 (day 1, 15, a total of 28 days).
  Repeat the cycle above until progression or intolerance of toxicity.
  Interventions: Drug: Sequential Treatment

INTERVENTIONS:
Drug: Sequential Treatment — One cycle of the treatment lasts for 56 days. Patients will receive chemotherapy based on Nab-paclitaxel Plus Gemcitabine and modified Folfirinox in sequence order. The cycle will repeat until progression or intolerance of toxicity.
  Other Names: Sequential Treatment With AG and Modified Folfirinox

SUMMARY:
The prognosis of pancreatic cancer is extremely poor. Current guidelines recommend Nab-paclitaxel, Gemcitabine and modified Folfirinox as the first-line chemotherapeutic regimen. Studies have shown that sequential chemotherapeutic regimen can effectively delay the drug resistance and improve the effect of chemotherapy. Here investigators intend to assess the effect of sequential treatment with Nab-paclitaxel plus Gemcitabine and modified Folfirinox on metastatic pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
Investigators chose metastatic pancreatic adenocarcinoma patients who can't meet surgical criteria. The planned treatment was given to the participants after enrollment. Objective remission rate, disease control rate, tumor size, progression-free survival, overall survival, drugs related side effects and other endpoints events were recorded and analyzed, to assess the sequential treatment with Nab-paclitaxel plus Gemcitabine and modified Folfirinox could or couldn't effectively control the progress of metastatic pancreatic adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically diagnosed metastatic pancreatic adenocarcinoma (excluding islet cell tumor) that can be measured according to RECIST criteria.
2. Without Radiotherapy, surgery, chemotherapy or experimental treatment for metastatic pancreatic cancer. Previous use of 5-FU or gemcitabine as a radiosensitizer in adjuvant therapy is allowed, but it should be taken at least 6 months ago and no residual toxicity. Patients receiving cytotoxic doses of gemcitabine or any other chemotherapy in adjuvant therapy are not eligible for this study.
3. ECOG score 0-1 points.
4. The first diagnosis time of metastatic pancreatic cancer should be within 6 weeks of the initial of treatment. Note: This interval is calculated from the date of final assessment of the confirmed pancreatic cancer metastasis.
5. No jaundice symptoms before treatment. Pain should be stable, and no need to adjust analgesic treatment. Patients with obvious or symptomatic ascites should be drained before treatment.
6. With enough blood cell counts during the screening period(less than 14 days before the treatment): 1) The absolute count of neutrophils(ANC) is more than 1.5 ×10^9/L; 2) Platelet count was greater than 100,000/mm^3 (100 x10^9/L); 3).

   Hemoglobin (Hgb) is more than 9 g/dL.
7. With normal blood biochemical parameters during the screening period(less than 14 days before the treatment): 1). AST (SGOT), ALT (SGPT) <2.5*ULN, if there is obvious liver metastasis, it is allowed to <5*ULN. 2). Total bilirubin is less than ULN. 3). Serum creatinine is within the normal limit, or the serum creatinine level is higher or lower than the normal value of the body, but the calculated clearance rate is more than 60 mL/min/1.73 m^2. If creatinine clearance is used, the actual body weight should be used to calculate creatinine clearance (for example, the Cockroft-Gault formula). Patients with body mass index (BMI) >30 kg/m^2 should use fat free body weight.
8. Acceptable coagulation test results (less than 14 days before treatment): prothrombin time (PT) and partial thromboplastin time (PPT) were within the normal limit (+15%).
9. With no clinically significant abnormal urine analysis (less than 14 days before treatment).
10. Male or non pregnant and non lactating women aged 18 or above who signed the informed consent.
11. Patients were informed of the nature of the study and agreed to participate in the study, and informed consent was signed before participating in any research-related activities.

Exclusion Criteria:

1. With brain metastases.
2. Only locally progressive diseases.
3. Serum albumin level decreased by more than 20% within 72 hours of first days before screening visit to first cycle.
4. With a history of malignancies (including chronic leukemia) over the past 5 years. Patients with previous history of carcinoma in situ or basal cell or squamous cell carcinoma can be included. Patients with other malignancies who have been cured by surgery or surgery plus radiotherapy alone and remain disease-free for at least five years are also eligible.
5. Suffering from active or uncontrollable bacterial, viral or fungal infections requiring systemic treatment.
6. Known HIV infection, and/or active hepatitis B virus or hepatitis C virus infection (for patients with history of HBV or HCV infection, should be discussed with researchers).
7. Major surgeries were performed within 4 weeks of the first day of treatment in this study (i.e. non-removal of organs for diagnostic biopsy).
8. Myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass grafting, New York Heart Association (NYHA) grade III-IV heart failure, uncontrolled hypertension, clinically significant arrhythmias or electrocardiographic (ECG) abnormalities, cerebrovascular accidents, transient ischemic attacks, epileptic seizures or clinically significant arrhythmia or abnormal electrocardiogram (ECG) history within 6 months before treatment.
9. With history of allergy or hypersensitivity of any research drug or its adjunct.The patient presents the events outlined in the "Contraindications or Special Warnings and Cautions" section of the product or control drug prescription information.
10. With history of connective tissue diseases (such as lupus, scleroderma, nodular arteritis).
11. With history of interstitial pneumonia, slow progressive dyspnea, dry cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, allergic pneumonia, or multiple allergies.
12. Any condition that may impair patient safety or integrity of research data, including serious medical risk factors, medical events, laboratory abnormalities, or mental illness.
13. Patients entering any other clinical study, testing for an intervention drug, or may interfere with the evaluation of this study procedure.
14. Patients are unwilling or unable to follow the research procedure or plan to take 7 or more consecutive days off during the study period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Up to approximately 60 months
  The time of initial response until documented tumor progression.

SECONDARY OUTCOMES:
Overall survival | Up to approximately 60 months
  The time of initial response until documented patient death.
Objective response rate | Up to approximately 60 months
  Percentage of people does not get worse for a period of time after diagnosis
Disease control rate | Up to approximately 60 months
  Percentage of patients whose cancer doesn't progress after treatment
Carbohydrate antigen 19-9 | Up to approximately 60 months
  Serum Carbohydrate antigen 19-9 level
EORTC QLQ - PAN26 | Up to approximately 60 months
  Assessed by the European Organization for Research and Treatment of Cancer Quality of Life-pancreatic cancer 26 score(EORTC QLQ - PAN26)
Common Toxicity Criteria for Adverse Effects | Up to approximately 60 months
  According to Common Toxicity Criteria for Adverse Effects version 4

CONTACTS AND LOCATIONS:
Locations (1):
- The second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided